CLINICAL TRIAL: NCT03728257
Title: Lung Transplant G0 (LTGO): Improving Self-Management of Exercise After Lung Transplantation
Acronym: LTGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Annette DeVito Dabbs, PhD, RN, Professor and Chairman, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19020357; 1R01NR017196-01A1 (NIH)
Record Dates: First submitted 2018-10-21; First posted 2018-11-02 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Exercise; Lung Transplantation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: There will be two groups. The research study that will compare two methods of self-managing exercise after receiving a lung transplant. These methods are a home-based exercise program plus self-monitoring or self-monitoring alone. The investigator would also like to collect information about the patients health and ability to exercise, and the amount of physical activity the participants do per day. The length of the study will be 6 months.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LTGO-Home Based Exercise (Experimental): The lung transplant recipient will receive LTGO- Home Based Exercise, a behavioral exercise intervention that consists of in-home exercise training integrated with behavioral coaching using tele-rehabilitation.
  Interventions: Behavioral: LTGO-Home Based Exercise
- Enhanced Usual Care (Active Comparator): Enhanced Usual Care (EUC) will involve delivery of monthly newsletters (6 newsletters) on the topics of post-lung transplant management, including food safety, environmental health, flu, mental health, etc. and the provision of a self-monitoring device.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: LTGO-Home Based Exercise — The LTGO intervention consists of two phases: Phase 1. Intensive home-based exercise training and behavioral coaching via a telerehabilitation platform, Versatile and Integrated System for Tele-Rehabilitation (VISYTER)/two-way video communication system. Interactive intervention sessions will be delivered to the home via real time video conferencing (up to 12 sessions and a behavioral contract plan to prepare for phase 2); and Phase 2. Transition to self-management. Three telephone sessions (3 monthly counseling sessions) will be delivered over 12 weeks to provide behavioral coaching and exercise reinforcement
  Arms: LTGO-Home Based Exercise
Behavioral: Enhanced Usual Care — Enhanced Usual Care (EUC) will involve delivery of monthly newsletters (6 newsletters) on the topics of post-lung transplant management, including food safety, environmental health, flu, mental health, etc. and the provision of a self-monitoring device.
  Arms: Enhanced Usual Care

SUMMARY:
Estimated costs, from thirty days prior to lung transplant up through six months post surgery, exceed 1 million dollars per patient and routine medical costs average approximately fifty thousand dollars per year thereafter. Prior to transplant, lung transplant recipients self restrict activity due to severe respiratory limitations, resulting in reduced muscle mass and qualitative changes in large skeletal muscles. After transplant, despite improved lung function, studies consistently report that lung recipients fail to reach predicted physical function and physical activity. Nearly seventy percent are at risk of developing hypertension within the first five years due to side effects of immunosuppression and an inactive lifestyle worsens this risk. Consequently, full benefits of transplant may not be achieved. Few studies have tested ways to engage lung recipients in self management of exercise and adopt an active lifestyle. Lung Transplant Go LTGO is a behavioral exercise intervention that provides individualized exercise training integrated with behavioral coaching delivered in the recipient's home. Exercise training will focus on assisting lung recipients to learn and practice exercises to reverse muscle conditioning. Behavioral coaching will assist them to develop the skills to self manage physical activity in daily life and maintain this as a sustained habit using strategies that include incremental goal setting, self-monitoring, feedback and problem solving.

DETAILED DESCRIPTION:
This is a two-group randomized controlled trial (RCT) comparing LTGO to enhanced usual care (EUC). Based on estimations using a published RCT, effect sizes measured by Cohen's d ranged from 0.64 to 1.45 across outcome variables (i.e., 0.64 for physical function; 0.73-0.99 for physical activity; and 1.19 and1.45 for systolic and diastolic BP with 80% power, α=0.05). With a final sample of 80 subjects (40 per group) we will have 80% power to detect an effect size as small as 0.64 (α=0.05, two-tailed) from independent sample t-test for measures of physical function, physical activity and hypertension onset/control. Recruiting and randomizing 112 individuals (56 in LTGO & 56 in EUC) will allow for up to 30% attrition. Participants will be randomized to LTGO or EUC (1:1). The biostatistician will randomize participants using a blocked randomization scheme, stratified by sex (male vs. female) and length of hospital stay (≤2 wks vs.>2 wks). The block size (2 or 4) will be randomly selected to prevent prediction of group assignment. An "intention-to-treat" (ITT) approach will be used. All subjects will be analyzed in the group to which they were randomly assigned, regardless of adherence to the protocol, treatment received, and/or withdrawal from the protocol. Endorsed by international regulatory guidelines, the ITT approach is widely used in RCT because it minimizes the potential for the introduction of biases into data analysis and maintains prognostic balance generated from original random treatment allocation. Although the ITT approach is recommended for efficacy analysis in RCTs, the sensitivity of the results assumes that ITT will be explored using information collected regarding fidelity and dosage (e.g., number of sessions completed).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

  ->4 weeks after the participant had lung transplant surgery
* Discharged from the hospital after your lung transplant surgery
* MD report of difficulty walking ¼ mile or climbing 10 steps without resting
* Medical monitor approves patient eligibility for participation

Exclusion Criteria:

* concurrent participation in a formal exercise program, e.g., pulmonary rehabilitation, during the active eligible study period with no plans to stop formal exercise
* having other chronic conditions that may severely limit participation in exercise training, i.e., cardiac, musculoskeletal or cognitive impairments
* does not have home internet or smart device with Bluetooth capabilities
* medical issue precluding participation
* declining to be asked screening questions, or declining an introduction to the research team to hear about research
* greater than 18 months post-transplant hospital discharge (time/scheduling delays, transportation issues, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annette DeVito Dabbs, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, School of Nursing, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hergenroeder AL, Willey B, Vendetti M, Dabbs AD. Exercise Progression Protocol for Lung Transplant GO: A Multicomponent Telerehab Exercise Intervention for Patients After Lung Transplantation. Cardiopulm Phys Ther J. 2023 Jan;34(1):2-12. doi: 10.1097/CPT.0000000000000203. Epub 2022 Mar 23. No abstract available. PMID 36644217
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853
- [Derived] Moon SJE, Dabbs AD, Hergenroeder AL, Vendetti ML, Jones KB, Willey BM, Morrell MR, Imes CC. Considerations for assessing physical function and physical activity in clinical trials during the COVID-19 pandemic. Contemp Clin Trials. 2021 Jun;105:106407. doi: 10.1016/j.cct.2021.106407. Epub 2021 Apr 20. PMID 33887443
- See also: Exercise Progression Protocol for LTGO — https://pubmed.ncbi.nlm.nih.gov/36644217/

RESULTS

PARTICIPANT FLOW:
Groups:
- LTGO-Home Based Exercise: The lung transplant recipient will receive LTGO- Home Based Exercise, a behavioral exercise intervention that consists of in-home exercise training integrated with behavioral coaching using tele-rehabilitation.
  LTGO-Home Based Exercise: The LTGO intervention consists of two phases: Phase 1.
  Intensive home-based exercise training and behavioral coaching via a telerehabilitation platform, VISYTER (Versatile and Integrated System for Tele-Rehabilitation)/two-way video communication system. Interactive intervention sessions will be delivered to the home via real time video conferencing (up to 12 sessions and a behavioral contract plan to prepare for phase 2); and Phase 2. Transition to self-management. Three telephone sessions (3 monthly counseling sessions) will be delivered over 12 weeks to provide behavioral coaching and exercise reinforcement
Period: Overall Study
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Started | 44 | 44
Completed | 41 | 44
Not Completed | 3 | 0
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.89 (14.01) | 57.93 (11.79) | 56.41 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex as documented in the electronic health record.
  Participants
    Female | 21 | 19 | 40
    Male | 23 | 25 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 42 | 42 | 84
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 36 | 42 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Average steps per day [Mean (Standard Deviation); unit: Average steps per day] — Average steps per day calculated by FitBit step tracker (FitBit) worn for 14 day periods at baseline. Minimum = 0, no upper limit. Higher scores mean a better outcome.
  Average steps per day | 3169.62 (2841.43) | 3507.14 (2535.84) | 3338.16 (2682.20)
Berg Balance [Mean (Standard Deviation); unit: units on a scale] — Balance was measured using the Berg Balance Score.This scale tests ability to handle tasks that require balance (e.g., sitting to standing, placing alternate foot on stool.) Minimum = 0, upper limit = 56. Higher scores indicate a better outcome.
  units on a scale | 53.69 (2.76) | 52.71 (4.30) | 53.21 (3.62)
Lower body strength [Mean (Standard Deviation); unit: Repetitions] — Lower body strength was measured with the 30-Second Chair-Stand Test. The participant will be instructed to: 1) sit in the middle of a chair (17 inch height, with a straight back without armrests); 2) place hands on the opposite shoulder crossed at the wrists; 3) keep feet flat on the floor and back straight. On "Go," the participant will be asked to rise to a full standing position, sit down on the chair and repeat this move for 30 seconds. Minimum score =0 with no upper limit. More repetitions indicate better outcome
  Repetitions | 9.64 (2.89) | 9.78 (3.57) | 9.70 (3.21)
Respiratory-related quality of life St George Respiratory Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Respiratory-related quality of life was measured with the St. George Respiratory Questionnaire (SGRQ). The SGRQ is a 50-item self-report measure that assesses symptoms and activities that cause or are limited by breathlessness. Minimum score = 0 with 100 upper limit. Higher scores indicate worse outcomes
  units on a scale | 31.65 (18.86) | 31.16 (19.89) | 31.40 (19.27)
Minutes per day in Moderate and Vigorous Physical Activity [Mean (Standard Deviation); unit: Minutes per day] — The number of minutes spent in moderate and vigorous physical activity per day was measured using the Actigraph Activity Tracker, an accelerometer to monitor physical activity. The device provides tri-axial vector data in activity units, metabolic equivalent tasks (METs), or kilocalories. The participant will wear the Actigraph for 7 days (starting the following day) during waking hours (≥10 hours of wear/day). Minutes spent in moderate and vigorous physical activity (MVPA) is summed for MVPA minutes/day. Minimum score = 0 with no upper limit. Higher scores indicate better outcomes
  Minutes per day | 11.5 (13.43) | 9.26 (9.35) | 10.12 (11.02)

OUTCOME MEASURES:

1. Primary Outcome: Physical Function- Walking: Change in Average Steps Per Day at Month 3
Description: Walking was measured as the change in average steps per day calculated by FitBit worn for periods at baseline and 3 months. Minimum = 0, no upper limit. Higher scores mean a better outcome. Change = (3 month score minus baseline score).
Time Frame: Baseline and 3 months
Population: Intent to Treat population (all participants randomized to LTGO or EUC). Compare difference between groups in change of average steps per day between baseline and 3 months.
Measure: Mean (Standard Deviation); unit: average steps per day
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 44 | 44
average steps per day | 460 (3410) | 352 (2470)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in average steps per day between baseline and 3 months was compared between the two groups; p = 0.8793, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

2. Primary Outcome: Physical Function- Walking: Change in Average Steps Per Day at Month 6
Description: Walking was measured as the change in average steps per day calculated by FitBit worn for periods at baseline and 6 months. Minimum = 0, no upper limit. Higher scores indicate a better outcome. Change = (6 month score minus baseline score).
Time Frame: Baseline and 6 months
Population: Intent to Treat population (all surviving participants randomized to LTGO or EUC). Compare difference between groups in change of average steps per day between baseline and 6 months.
Measure: Mean (Standard Deviation); unit: average steps per day
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 41 | 44
average steps per day | 445 (2310) | 405 (3570)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in average steps per day between baseline and 6 months was compared between the two groups; p = 0.9597, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

3. Primary Outcome: Physical Function- Balance: Change in Berg Balance at Month 3
Description: Balance was measured as the change in Berg Balance Score at baseline and 3 months. This scale tests ability to handle tasks that require balance (e.g., sitting to standing, placing alternate foot on stool.) Minimum = 0, upper limit = 56.
  Higher scores indicate a better outcome. Change = (3 month score minus baseline score).
Time Frame: Baseline and 3 months.
Population: Intent to Treat population (all participants randomized to LTGO or EUC). Compare difference between groups in change of Berg Balance between baseline and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 44 | 44
units on a scale | 0.48 (1.96) | 0.67 (1.67)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in Berg balance between baseline and 3 months was compared between the two groups; p = 0.30, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

4. Primary Outcome: Physical Function- Balance: Change From Baseline to 6 Months
Description: Balance was measured as the change in Berg Balance Score at baseline and 6 months. This scale tests ability to handle tasks that require balance (e.g., sitting to standing, placing alternate foot on stool.) Minimum = 0, upper limit = 56.
  Higher scores indicate a better outcome. Change = (6 month score minus baseline score).
Time Frame: Baseline and 6 months
Population: Intent to Treat population (all surviving participants randomized to LTGO or EUC). Compare difference between groups in change of Berg Balance between baseline and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 41 | 44
units on a scale | 1.71 (3.29) | 0.74 (1.73)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in Berg balance between baseline and 3 months was compared between the two groups; p = 0.81, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

5. Primary Outcome: Physical Function-Lower Body Strength: Change From Baseline to 3 Months
Description: Lower body strength was measured as the change in 30-Second Chair Stand Test at baseline and 3 months. The participant will be instructed to: 1) sit in the middle of a chair (17 inch height, with a straight back without armrests); 2) place hands on the opposite shoulder crossed at the wrists; 3) keep feet flat on the floor and back straight. On "Go," the participant will be asked to rise to a full standing position, sit down on the chair and repeat this move for 30 seconds. Minimum score =0 with no upper limit. More repetitions indicate better outcome. Change = (3 month score minus baseline score).
Time Frame: Baseline and 3 months.
Population: Intent to Treat population (all participants randomized to LTGO or EUC). Compare difference between groups in change of 30-Second Chair Stand Test between baseline and 3 months.
Measure: Mean (Standard Deviation); unit: repetitiions
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 44 | 44
repetitiions | 0.964 (2.03) | 0.314 (2.18)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in 30 Second Sit-to-Stand Test between baseline and 3 months was compared between the two groups; p = 0.2262, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance is p < 0.05

6. Primary Outcome: Physical Function-Lower Body Strength: Change From Baseline to 6 Months
Description: Lower body strength was measured as the change in 30-Second Chair Stand Test at baseline and 6 months. The participant will be instructed to: 1) sit in the middle of a chair (17 inch height, with a straight back without armrests); 2) place hands on the opposite shoulder crossed at the wrists; 3) keep feet flat on the floor and back straight. On "Go," the participant will be asked to rise to a full standing position, sit down on the chair and repeat this move for 30 seconds. Minimum score = 0 with no upper limit. More repetitions indicate better outcome. Change = (6 month score minus baseline score).
Time Frame: Baseline and 6 months.
Population: Intent to Treat population (all surviving participants randomized to LTGO or EUC). Compare difference between groups in change of 30-Second Chair Stand Test between baseline and 6 months.
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 41 | 44
repetitions | 1.5 (2.53) | 1.11 (3.29)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in 30 Second Sit-to-Stand Test between baseline and 6 months was compared between the two groups; p = 0.59, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

7. Primary Outcome: Physical Function- Respiratory-related Quality of Life Change From Baseline to 3 Months.
Description: Respiratory-related quality of life was measured as the change in the St. George Respiratory Questionnaire (SGRQ) at baseline and 3 months. The SGRQ is a 50-item self-report measure that assesses symptoms and activities that cause or are limited by breathlessness. Minimum score = 0 with 100 upper limit. Higher scores indicate worse outcomes. Change = (3 month score minus baseline score).
Time Frame: Baseline and 3 months.
Population: Intent to Treat population (all participants randomized to LTGO or EUC). Compare difference between groups in change of SGRQ between baseline and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 44 | 44
units on a scale | -4.64 (9.29) | -6.45 (11.56)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in SGRQ between baseline and 3 months was compared between the two groups; p = 0.26, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

8. Primary Outcome: Physical Function- Respiratory-related Quality of Life: Change From Baseline to 6 Months.
Description: Respiratory-related quality of life was measured as the change in the St. George Respiratory Questionnaire (SGRQ) at baseline and 6 months. The SGRQ is a 50-item self-report measure that assesses symptoms and activities that cause or are limited by breathlessness. Minimum score = 0 with 100 upper limit. Higher scores indicate worse outcomes. Change = (6 month score minus baseline score).
Time Frame: Baseline and 6 months
Population: Intent to Treat population (all surviving participants randomized to LTGO or EUC). Compare difference between groups in change of respiratory-related quality of life between baseline and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 41 | 44
units on a scale | -6.33 (11.26) | -6.83 (8.38)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in SGRQ between baseline and 6 months was compared between the two groups; p = 0.78, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

9. Primary Outcome: Physical Activity-Minutes of Moderate to Vigorous Physical Activity Per Day: Change From Baseline to 3 Months.
Description: The number of minutes spent in moderate and vigorous physical activity per day was measured using the Actigraph, an accelerometer to monitor physical activity. The device provides tri-axial vector data in activity units, metabolic equivalent tasks (METs), or kilocalories. The participant will wear the Actigraph for 7 days (starting the following day) during waking hours (≥10 hours of wear/day). Minutes spent in moderate and vigorous physical activity (MVPA) is summed for MVPA minutes/day. Minimum score = 0 with no upper limit. Higher scores indicate better outcomes. Change = (3 month score minus baseline score).
Time Frame: Baseline and 3 months.
Population: Intent to Treat population (all participants randomized to LTGO or EUC). Compare difference between groups in change of MVPA between baseline and 3 months.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 44 | 44
minutes per day | 2.18 (7.37) | 1.17 (13.0)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in MVPA between baseline and 3 months was compared between the two groups; p = 0.7073, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

10. Primary Outcome: Physical Activity-Moderate to Vigorous Physical Activity Per Day: Change From Baseline to 6 Months.
Description: The number of minutes spent in moderate and vigorous physical activity per day was measured using the Actigraph, an accelerometer to monitor physical activity. The device provides tri-axial vector data in activity units, metabolic equivalent tasks (METs), or kilocalories. The participant will wear the Actigraph for 7 days (starting the following day) during waking hours (≥10 hours of wear/day). Minutes spent in moderate and vigorous physical activity (MVPA) is summed for MVPA minutes/day. Minimum score = 0 with no upper limit. Higher scores indicate better outcomes. Change = (6 month score minus baseline score).
Time Frame: Baseline and 6 months.
Population: Intent to Treat population (all surviving participants randomized to LTGO or EUC). Compare difference between groups in change of MVPA between baseline and 6 months.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 41 | 44
minutes per day | 2.38 (9.99) | 6.53 (21.6)
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in MVPA between baseline and 6 months was compared between the two groups; p = 0.313, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance p < 0.05

11. Secondary Outcome: Blood Pressure Control-Change From Baseline to 3months
Description: Blood pressure control was measured as change in stage of hypertension. Systolic and diastolic blood pressure was assessed, then categorized from 1 (normal) to 4 (stage 3) according to the standard categories for hypertension. Change was calculated as stage at 3 months minus stage at baseline -3 to +3. Difference reported as the count of participants whose BP stage remained the same or improved between baseline and 3 months. A higher count indicates better outcome.
Time Frame: Baseline and 3 months
Population: Intent to Treat population (all participants randomized to LTGO or EUC). Compare difference between groups in counts of participants with the same or improved stage of hypertension between baseline and 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 44 | 44
Participants | 30 | 31
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in count of participants with the same or improved stage of hypertension between baseline and 6 months; p = 0.91, Chi-squared — a priori threshold for statistical significance p < 0.05

12. Secondary Outcome: Blood Pressure Control-Change From Baseline to 6 Months
Description: Blood pressure control was measured as change in stage of hypertension. Systolic and diastolic blood pressure was assessed, then categorized from 1 (normal) to 4 (stage 3) according to the standard categories for hypertension. Change was calculated as stage at 6 months minus stage at baseline -3 to +3. Difference reported as the count of participants whose BP stage remained the same or improved between baseline and 6 months. A higher count indicates better outcome.
Time Frame: Baseline and 6 months.
Population: Intent to Treat population (all surviving participants randomized to LTGO or EUC). Compare difference between groups in counts of participants with the same or improved stage of hypertension between baseline and 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
Number analyzed (Participants) | 41 | 44
Participants | 30 | 24
Statistical Analysis 1: Comparison: LTGO-Home Based Exercise vs Enhanced Usual Care; Test type: Superiority — Change in count of participants with the same or improved stage of hypertension between baseline and 6 months; p = 0.72, Chi-squared — a priori threshold of statistical significance p < 0.05

ADVERSE EVENTS:
Time Frame: up to 6 months
Description: Per our data safety protocol of the University of Pittsburgh Institutional Review Board (IRB), the definitions of adverse events and or serious adverse events were limited to unanticipated events. Since mortality is an expected event in this population, the causes were reviewed according to our protocol and deemed anticipated and unrelated to participation in this study.
Arm/Group | LTGO-Home Based Exercise | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 3/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT03728257/Prot_SAP_000.pdf